CLINICAL TRIAL: NCT05296395
Title: Impact of Lp299v on Vascular Aging in Healthy Adults
Brief Title: Vascular Aging and Lp299v Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Michael E. Widlansky, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PRO43157
Record Dates: First submitted 2022-03-15; First posted 2022-03-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Vascular Aging
Keywords: Endothelial Function; Microbiome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lp299v (Experimental): Subjects will consume 20 billion colony forming units of Lp299v (1 serving of GoodBelly fermented oat drink) once daily for 6 weeks
  Interventions: Other: Lactobacillus Plantarum 299v in fermented oat drink
- Heat-killed placebo control (Placebo Comparator): Subjects will consume 1 serving of GoodBelly fermented oat drink that has been treated to heat kill all Lp299v once daily for 6 weeks
  Interventions: Other: Heat-Killed Placebo control fermented drink

INTERVENTIONS:
Other: Lactobacillus Plantarum 299v in fermented oat drink — The intervention is a probiotic lactobacillus that is contained in food products in the US
  Other Names: GoodBelly StraighShot
  Arms: Lp299v
Other: Heat-Killed Placebo control fermented drink — The intervention is the GoodBelly StraightShort that has been treated to heat kill all Lp299v
  Arms: Heat-killed placebo control

SUMMARY:
Emerging data suggest the gut microbiota regulates multiple mechanisms related to vascular aging, but no intervention targeting the gut microbiota has been tested in older adults without cardiovascular risk factors or cardiovascular disease. Early human data suggest an increase in potentially pathological gut metabolites such as trimethylamine-N-oxide (TMAO) are associated with older age, increased vascular stiffness, increased oxidative stress, and reduced nitric oxide (NO) bioavailability as evidenced by impaired endothelium-dependent vasodilation. Based on this data, the investigators hypothesize that supplementation with Lp299v will reverse human vascular aging in healthy older adults free of known traditional cardiovascular risk factors.

DETAILED DESCRIPTION:
Multiple lines of evidence suggest that aging results in significant changes in the composition and metabolism of the gut microbiota that accelerate mechanisms responsible for vascular aging. Recent work established cross-sectional associations between phenotypically older vasculature (with increased vascular stiffness and impaired brachial endothelium-dependent vasodilation) and age-related alterations on the composition of the gut microbiota and metabolites that are derived from microbial metabolism such as TMAO (trimethylamine-N-oxide), nicotinamide, tryptophan, and purines. Animal data also suggests short-chain fatty acids favorably impact endothelium-dependent vasodilation. SCFAs exert a direct anti-inflammatory effect on mononuclear cells and increase glucagon-like protein 1 (GLP-1) production which activates endothelial nitric oxide synthase (eNOS) and increases NO levels. Taken together, these data suggest aging-related changes in the gut microbiota could adversely affect vascular health through multiple mechanisms, even in the absence of concomitant cardiovascular risk factors.

Six weeks of Lp299v supplementation in 36 otherwise healthy smokers reduced systemic inflammation, as evidenced by reductions in leptin (an adipokine that stimulates IL-6 production) and IL-6 levels, reduced monocyte adhesion to endothelial cells, and reduced circulating fibrinogen levels (elevated in the setting of inflammation). In addition, Lp299v supplementation reduced oxidative stress based on reduced urinary F2-isoprostanes and had a modest lowering effect on systolic blood pressure.

The investigators will recruit 20 healthy older adults (10 men, 10 women ages 50 or older) without traditional cardiac risk factors or prevalent cardiovascular disease and randomize subjects into a 6-week, double-blind, randomized, placebo-controlled clinical trial of Lp299v supplementation. Measurements of micro-and macrovascular function, systemic inflammation, and stool microbiota composition will be made.

ELIGIBILITY:
Inclusion Criteria:

* Ages 50-99 years
* For women: 12 months or more since last menstruation

Exclusion Criteria:

* Systolic Blood Pressure ≥ 130 mmHg or Diastolic BP ≥ 80mmHg
* Currently taking pharmacological therapies for hypertension, dyslipidemia, or glucose control
* Diabetes (type 1 or 2) or glycosylated hemoglobin ≥ 5/7%
* LDL Cholesterol > 160 mg/dL or Total Cholesterol > 200 mg/dL
* Cigarette use within 3 years of enrollment
* Average of > 7500 steps per day as measured during screening period
* Received probiotics, prebiotics, and/or antibiotics within six weeks of enrollment
* History of chronic renal insufficiency, liver dysfunction, or cancer besides non-melanoma skin carcinomas or localized prostate cancer requiring systemic treatment within 3 years of enrollment
* History of inflammatory rheumatic diseases known to increase atherosclerotic cardiovascular risk (e.g. rheumatoid arthritis, systemic lupus erythematosus)
* Known history of cognitive impairment or inability to follow study procedures
* GI tract illnesses such as short gut syndrome, inflammatory bowel disease, or an ileostomy
* Daily alcohol use

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2027-09-22 (Estimated)

PRIMARY OUTCOMES:
Brachial Artery Flow Mediated Dilation (FMD% | 6 weeks
  This is a measurement of endothelial function in the brachial artery

SECONDARY OUTCOMES:
Nitroglycerin-Mediated Vasodilation of the brachial artery (NMD) | 6 weeks
  Measurement of vascular smooth muscle reactivity
Hyperemic Flow Velocity | 6 weeks
  Measurement of microvascular endothelial function
Carotid-Femoral Pulse Wave Velocity (cfPWV) | 6 weeks
  Measurement of vascular stiffness
Stool microbiota alpha diversity | 6 weeks
  Diversity of bacterial species in the individual microbiome
Stool microbiota beta diversity | 6 weeks
  Differences in bacterial composition between intervention arms
Brachial Artery Resting Diameter | 6 weeks
  resting diameter of the brachial artery - representative of resting vascular tone

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Widlansky, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
All data that are relevant to publication of the results of this work
Supporting Information: Study Protocol, ICF
Time Frame: Within 1 year of completion of publication of study.
Access Criteria: Data will be available to qualified investigators.

REFERENCES:
- [Background] Claesson MJ, Cusack S, O'Sullivan O, Greene-Diniz R, de Weerd H, Flannery E, Marchesi JR, Falush D, Dinan T, Fitzgerald G, Stanton C, van Sinderen D, O'Connor M, Harnedy N, O'Connor K, Henry C, O'Mahony D, Fitzgerald AP, Shanahan F, Twomey C, Hill C, Ross RP, O'Toole PW. Composition, variability, and temporal stability of the intestinal microbiota of the elderly. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4586-91. doi: 10.1073/pnas.1000097107. Epub 2010 Jun 22. PMID 20571116
- [Background] Hebuterne X. Gut changes attributed to ageing: effects on intestinal microflora. Curr Opin Clin Nutr Metab Care. 2003 Jan;6(1):49-54. doi: 10.1097/00075197-200301000-00008. PMID 12496680
- [Background] Menni C, Lin C, Cecelja M, Mangino M, Matey-Hernandez ML, Keehn L, Mohney RP, Steves CJ, Spector TD, Kuo CF, Chowienczyk P, Valdes AM. Gut microbial diversity is associated with lower arterial stiffness in women. Eur Heart J. 2018 Jul 1;39(25):2390-2397. doi: 10.1093/eurheartj/ehy226. PMID 29750272
- [Background] Schirmer M, Smeekens SP, Vlamakis H, Jaeger M, Oosting M, Franzosa EA, Ter Horst R, Jansen T, Jacobs L, Bonder MJ, Kurilshikov A, Fu J, Joosten LAB, Zhernakova A, Huttenhower C, Wijmenga C, Netea MG, Xavier RJ. Linking the Human Gut Microbiome to Inflammatory Cytokine Production Capacity. Cell. 2016 Nov 3;167(4):1125-1136.e8. doi: 10.1016/j.cell.2016.10.020. PMID 27814509
- [Background] Brunt VE, Gioscia-Ryan RA, Richey JJ, Zigler MC, Cuevas LM, Gonzalez A, Vazquez-Baeza Y, Battson ML, Smithson AT, Gilley AD, Ackermann G, Neilson AP, Weir T, Davy KP, Knight R, Seals DR. Suppression of the gut microbiome ameliorates age-related arterial dysfunction and oxidative stress in mice. J Physiol. 2019 May;597(9):2361-2378. doi: 10.1113/JP277336. Epub 2019 Feb 27. PMID 30714619
- [Background] Brunt VE, Gioscia-Ryan RA, Casso AG, VanDongen NS, Ziemba BP, Sapinsley ZJ, Richey JJ, Zigler MC, Neilson AP, Davy KP, Seals DR. Trimethylamine-N-Oxide Promotes Age-Related Vascular Oxidative Stress and Endothelial Dysfunction in Mice and Healthy Humans. Hypertension. 2020 Jul;76(1):101-112. doi: 10.1161/HYPERTENSIONAHA.120.14759. Epub 2020 Jun 10. PMID 32520619
- [Background] Ke Y, Li D, Zhao M, Liu C, Liu J, Zeng A, Shi X, Cheng S, Pan B, Zheng L, Hong H. Gut flora-dependent metabolite Trimethylamine-N-oxide accelerates endothelial cell senescence and vascular aging through oxidative stress. Free Radic Biol Med. 2018 Feb 20;116:88-100. doi: 10.1016/j.freeradbiomed.2018.01.007. Epub 2018 Jan 8. PMID 29325896
- [Background] Li T, Chen Y, Gua C, Li X. Elevated Circulating Trimethylamine N-Oxide Levels Contribute to Endothelial Dysfunction in Aged Rats through Vascular Inflammation and Oxidative Stress. Front Physiol. 2017 May 30;8:350. doi: 10.3389/fphys.2017.00350. eCollection 2017. PMID 28611682
- [Background] Brandsma E, Kloosterhuis NJ, Koster M, Dekker DC, Gijbels MJJ, van der Velden S, Rios-Morales M, van Faassen MJR, Loreti MG, de Bruin A, Fu J, Kuipers F, Bakker BM, Westerterp M, de Winther MPJ, Hofker MH, van de Sluis B, Koonen DPY. A Proinflammatory Gut Microbiota Increases Systemic Inflammation and Accelerates Atherosclerosis. Circ Res. 2019 Jan 4;124(1):94-100. doi: 10.1161/CIRCRESAHA.118.313234. PMID 30582442
- [Background] Schirmer M, Smeekens SP, Vlamakis H, Jaeger M, Oosting M, Franzosa EA, Horst RT, Jansen T, Jacobs L, Bonder MJ, Kurilshikov A, Fu J, Joosten LAB, Zhernakova A, Huttenhower C, Wijmenga C, Netea MG, Xavier RJ. Linking the Human Gut Microbiome to Inflammatory Cytokine Production Capacity. Cell. 2016 Dec 15;167(7):1897. doi: 10.1016/j.cell.2016.11.046. No abstract available. PMID 27984736
- [Background] Geva-Zatorsky N, Sefik E, Kua L, Pasman L, Tan TG, Ortiz-Lopez A, Yanortsang TB, Yang L, Jupp R, Mathis D, Benoist C, Kasper DL. Mining the Human Gut Microbiota for Immunomodulatory Organisms. Cell. 2017 Feb 23;168(5):928-943.e11. doi: 10.1016/j.cell.2017.01.022. Epub 2017 Feb 16. PMID 28215708
- [Background] Sharma R, Padwad Y. Probiotic bacteria as modulators of cellular senescence: emerging concepts and opportunities. Gut Microbes. 2020 May 3;11(3):335-349. doi: 10.1080/19490976.2019.1697148. Epub 2019 Dec 10. PMID 31818183
- [Background] Wu CS, Muthyala SDV, Klemashevich C, Ufondu AU, Menon R, Chen Z, Devaraj S, Jayaraman A, Sun Y. Age-dependent remodeling of gut microbiome and host serum metabolome in mice. Aging (Albany NY). 2021 Feb 17;13(5):6330-6345. doi: 10.18632/aging.202525. Epub 2021 Feb 17. PMID 33612480
- [Background] Natarajan N, Hori D, Flavahan S, Steppan J, Flavahan NA, Berkowitz DE, Pluznick JL. Microbial short chain fatty acid metabolites lower blood pressure via endothelial G protein-coupled receptor 41. Physiol Genomics. 2016 Nov 1;48(11):826-834. doi: 10.1152/physiolgenomics.00089.2016. Epub 2016 Sep 23. PMID 27664183
- [Background] Tolhurst G, Heffron H, Lam YS, Parker HE, Habib AM, Diakogiannaki E, Cameron J, Grosse J, Reimann F, Gribble FM. Short-chain fatty acids stimulate glucagon-like peptide-1 secretion via the G-protein-coupled receptor FFAR2. Diabetes. 2012 Feb;61(2):364-71. doi: 10.2337/db11-1019. Epub 2011 Dec 21. PMID 22190648
- [Background] Ding L, Zhang J. Glucagon-like peptide-1 activates endothelial nitric oxide synthase in human umbilical vein endothelial cells. Acta Pharmacol Sin. 2012 Jan;33(1):75-81. doi: 10.1038/aps.2011.149. Epub 2011 Nov 28. PMID 22120969
- [Background] Chai W, Dong Z, Wang N, Wang W, Tao L, Cao W, Liu Z. Glucagon-like peptide 1 recruits microvasculature and increases glucose use in muscle via a nitric oxide-dependent mechanism. Diabetes. 2012 Apr;61(4):888-96. doi: 10.2337/db11-1073. Epub 2012 Feb 22. PMID 22357961
- [Background] Tsiotra PC, Boutati E, Dimitriadis G, Raptis SA. High insulin and leptin increase resistin and inflammatory cytokine production from human mononuclear cells. Biomed Res Int. 2013;2013:487081. doi: 10.1155/2013/487081. Epub 2012 Dec 24. PMID 23484124
- [Background] Yang WH, Liu SC, Tsai CH, Fong YC, Wang SJ, Chang YS, Tang CH. Leptin induces IL-6 expression through OBRl receptor signaling pathway in human synovial fibroblasts. PLoS One. 2013 Sep 27;8(9):e75551. doi: 10.1371/journal.pone.0075551. eCollection 2013. PMID 24086566
- [Background] Tang CH, Lu DY, Yang RS, Tsai HY, Kao MC, Fu WM, Chen YF. Leptin-induced IL-6 production is mediated by leptin receptor, insulin receptor substrate-1, phosphatidylinositol 3-kinase, Akt, NF-kappaB, and p300 pathway in microglia. J Immunol. 2007 Jul 15;179(2):1292-302. doi: 10.4049/jimmunol.179.2.1292. PMID 17617622
- [Background] Tazawa R, Uchida K, Fujimaki H, Miyagi M, Inoue G, Sekiguchi H, Murata K, Takata K, Kawakubo A, Takaso M. Elevated leptin levels induce inflammation through IL-6 in skeletal muscle of aged female rats. BMC Musculoskelet Disord. 2019 May 10;20(1):199. doi: 10.1186/s12891-019-2581-5. PMID 31077169
- [Background] Naruszewicz M, Johansson ML, Zapolska-Downar D, Bukowska H. Effect of Lactobacillus plantarum 299v on cardiovascular disease risk factors in smokers. Am J Clin Nutr. 2002 Dec;76(6):1249-55. doi: 10.1093/ajcn/76.6.1249. PMID 12450890